CLINICAL TRIAL: NCT01947712
Title: Effect of Dark Chocolate on Endothelial Function and Oxidative Stress in Patients With Peripheral Vascular Disease.
Brief Title: Effect of Polyphenols on Peripheral Vascular Disease.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Violi, Full professor of Internal Medicine, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: C26A12BPZN; C26A12BPZN (Other: Sapienza University)
Record Dates: First submitted 2013-09-12; First posted 2013-09-20 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral arterial disease; Oxidative stress; Cocoa; polyphenols; NADPH oxidase
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- milk chocolate (Placebo Comparator): dosage form: orally given dosage:40 g milk chocolate (≤35% cocoa) frequency and duration: 40 g/day for one month
  Interventions: Dietary Supplement: milk chocolate with crossover to dark chocolate
- dark chocolate (Active Comparator): dosage form: orally given dosage:40 g dark chocolate (≥85% cocoa) frequency and duration: 40 g/day for one month
  Interventions: Dietary Supplement: dark chocolate with crossover to milk chocolate

INTERVENTIONS:
Dietary Supplement: dark chocolate with crossover to milk chocolate — 40 g/d of dark chocolate for 4 weeks followed by wash-out (1 week) and by 40 g/d of milk chocolate for 4 weeks
  Arms: dark chocolate
Dietary Supplement: milk chocolate with crossover to dark chocolate — 40 g/d of milk chocolate for 4 weeks followed by wash-out (1 week) and by 40 g/d of dark chocolate for 4 weeks.
  Arms: milk chocolate

SUMMARY:
Peripheral arterial disease (PAD) is a clinical setting characterized by an exceptionally high risk for cardiovascular events. Oxidative stress seems to play a role in impairing flow-mediated dilation (FMD) and contributing to atherosclerosis in patients with PAD. Cocoa seems to exert artery dilatation via oxidative stress inhibition.

OBJECTIVES: To investigate whether in PAD patients, dark chocolate elicits artery dilatation via down-regulation of NOX2, the catalytic core of NADPH oxidase.

DETAILED DESCRIPTION:
Atherosclerosis represents the major cause of worldwide death; it is a complex phenomenon that encompasses the intricate interplay of classic cardiovascular risk factors, oxidative stress and inflammation.

Peripheral artery disease (PAD) is a clinical setting that well represents the model of widespread atherosclerosis. PAD affects 20% of patients over the age of 75. Furthermore, PAD patients are at an exceptionally high risk for cardiovascular events and the majority will eventually die of a cardiac or cerebrovascular etiology.

Polyphenol could represent a novel therapeutic strategy to counteract atherosclerosis. During the last decades, a growing interest in polyphenols resulted from prospective and epidemiological studies that showed the beneficial effects of these substances on human health. In particular, polyphenols exert their beneficial effect by inhibition of NADPH oxidase (NOX2), an enzyme directly involved in atherosclerosis; thus, the activation of this enzyme leads to an enhanced production of oxidative stress and inflammatory processes.

The objective of this study is to evaluate the effect of polyphenols on oxidative stress and inflammation and on surrogate markers of atherosclerosis in PAD patients. Polyphenols, inhibiting NOX2-mediated oxidative stress and immune-mediated process, could represent a novel therapy to reduce the high risk of cardiovascular events in PAD.

ELIGIBILITY:
Inclusion Criteria:

Every PAD patient to be enrolled in the study had:

1. claudication (defined as leg pain on walking, disappearing within 10 minutes of standing, of presumed atherosclerotic origin) and
2. ankle/brachial index (ABI), that was assessed as ankle/arm systolic blood pressure ratio by Doppler ultrasonography <0.90 on the worst leg at rest.

Patients had to be in stable conditions without abrupt changes of ABI (>20%) in the last month before the enrolment.

Exclusion Criteria:

Subjects were excluded from the study if they had liver insufficiency, serious renal disorders (serum creatinine>2.8 mg/dL), acute stroke, acute myocardial infarction, deep venous thrombosis or if they were current smokers or were taking antioxidants.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
endothelial function assessed by flow mediated dilation (FMD) | 2 hours after (dark or milk) chocolate ingestion
endothelial function assessed by flow mediated dilation (FMD) | after 30 days of (dark or milk) chocolate ingestion

SECONDARY OUTCOMES:
Oxidative stress markers | 2 hours after (dark or milk) chocolate ingestion
  Oxidative stress markers: sNOX2dp, Isoprostanes, NOx
Maximal walking distance | 2 hours after (dark or milk) chocolate ingestion
Ankle Brachial Index (ABI) | 2 hours after (dark or milk) chocolate ingestion
Oxidative stress markers | after 30 days of (dark or milk) chocolate ingestion
  Oxidative stress markers: sNOX2dp, Isoprostanes, NOx
Maximal walking distance | after 30 days of (dark or milk) chocolate ingestion
Ankle Brachial Index (ABI) | after 30 days of (dark or milk) chocolate ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Violi, MD, Principal Investigator — Sapienza University
Locations (1):
- Sapienza University of Rome, I Clinica Medica, Research Tower, Rome, Italy

REFERENCES:
- [Background] Loffredo L, Carnevale R, Cangemi R, Angelico F, Augelletti T, Di Santo S, Calabrese CM, Della Volpe L, Pignatelli P, Perri L, Basili S, Violi F. NOX2 up-regulation is associated with artery dysfunction in patients with peripheral artery disease. Int J Cardiol. 2013 Apr 30;165(1):184-92. doi: 10.1016/j.ijcard.2012.01.069. Epub 2012 Feb 14. PMID 22336250
- [Background] Carnevale R, Loffredo L, Pignatelli P, Nocella C, Bartimoccia S, Di Santo S, Martino F, Catasca E, Perri L, Violi F. Dark chocolate inhibits platelet isoprostanes via NOX2 down-regulation in smokers. J Thromb Haemost. 2012 Jan;10(1):125-32. doi: 10.1111/j.1538-7836.2011.04558.x. PMID 22066819
- [Background] Loffredo L, Carnevale R, Perri L, Catasca E, Augelletti T, Cangemi R, Albanese F, Piccheri C, Nocella C, Pignatelli P, Violi F. NOX2-mediated arterial dysfunction in smokers: acute effect of dark chocolate. Heart. 2011 Nov;97(21):1776-81. doi: 10.1136/heartjnl-2011-300304. Epub 2011 Jul 31. PMID 21807659
- [Derived] Loffredo L, Perri L, Catasca E, Pignatelli P, Brancorsini M, Nocella C, De Falco E, Bartimoccia S, Frati G, Carnevale R, Violi F. Dark chocolate acutely improves walking autonomy in patients with peripheral artery disease. J Am Heart Assoc. 2014 Jul 2;3(4):e001072. doi: 10.1161/JAHA.114.001072. PMID 24990275